CLINICAL TRIAL: NCT04462276
Title: Thoracic RadiothErapy With Atezolizumab in Small Cell lUng canceR Extensive Disease: a Randomized, Open-label, Multicenter Phase II Study
Brief Title: Thoracic RadiothErapy With Atezolizumab in Small Cell lUng canceR Extensive Disease
Acronym: TREASURE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Collaborators: Thoraxklinik-Heidelberg gGmbH (Other); Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TREASURE
Record Dates: First submitted 2020-06-28; First posted 2020-07-08 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Small Cell Lung Cancer Extensive Stage; Thoracic Radiotherapy
Keywords: SCLC; thoracic radiotherapy; Atezolizumab
MeSH Terms: interventions — atezolizumab

STUDY DESIGN:
Intervention Model Description: Randomized, open label, multicenter, phase II trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: Atezolizumab + thoracic radiotherapy (Experimental): Atezolizumab at a fixed dose of 1,200 mg as an IV infusion, on day 1, to be repeated every 3 weeks (Q3W) Thoracic radiation therapy (TRT), 30 Gy in 10 fractions
  Interventions: Drug: Atezolizumab; Radiation: thoracic radiotherapy (TRT)
- Arm B: Atezolizumab (Experimental): Atezolizumab at a fixed dose of 1,200 mg as an IV infusion, on day 1, to be repeated every 3 weeks (Q3W)
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Atezolizumab — fixed dose of 1,200 mg as an IV infusion, on day 1, to be repeated every 3 weeks (Q3W)
Radiation: thoracic radiotherapy (TRT) — 30 Gy in 10 fractions
  Arms: Arm A: Atezolizumab + thoracic radiotherapy

SUMMARY:
This is a multicenter phase 2 clinical trial to investigate the treatment efficacy and feasibility of combining thoracic radiotherapy (TRT) with the IMpower133 regimen in the upfront treatment of ED SCLC patients. Patients with a response after induction therapy with carboplatin/etoposide and atezolizumab will be included into this study to subsequently receive atezolizumab maintenance therapy and will be randomized to receive TRT or not. This trial aims to i.) increase the efficacy of combined atezolizumab- and chemotherapy by adding radiotherapy and ii.) determine the safety and tolerability of the combination of chemotherapeutic, immunological and radiological treatment in the first-line setting of advanced SCLC, and iii.) to collect tumor tissue as well as blood and stool samples for separate biomarker research project.

ELIGIBILITY:
Inclusion Criteria:

1. Fully-informed written consent and locally required authorization (European Union [EU] Data Privacy Directive in the EU) obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations.
2. Age ≥ 18 years.
3. Histologically or cytologically confirmed ED SCLC as defined according to the Veterans Administration Lung Study Group staging system.
4. Measurable ED SCLC according to Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1. In cases of CR or PR without residual measurable disease after 4 cycles of induction therapy, patients may still be included. In such cases "No Evidence of Disease (NED)" should be reported in eCRF.
5. ECOG performance status score of 0 or 1 at screening
6. Any response after four cycles of standard chemo-immunotherapy (carboplatin, etoposide, atezolizumab) defined as CR/PR or thoracic SD with CR/PR of extrathoracic lesions as per RECIST 1.1
7. Thoracic treatment volume considered treatable using acceptable radiation fields as judged by a radiation oncologist
8. 28 ± 7 days between last administration of chemo-immunotherapy (carboplatin, etoposide, atezolizumab) and randomization.
9. Patients with a history of treated CNS metastases are eligible, if there is no ongoing requirement for corticosteroids as therapy for CNS disease. Before randomization, MRI of brain (with contrast, unless contraindicated) is recommended in subjects with suspected or known brain metastases, as per local standard., Patients with asymptomatic brain metastases that do not require local therapy with irradiation (whole brain irradiation) can be included. In ambiguous cases, consultation with the LKP or his/her delegate is advised.
10. No previous radiotherapy to lung and mediastinal lymph nodes within the past 5 years before the first dose of study drug.
11. Availability of pre-treatment tumor tissue specimen
12. The patient is willing and able to comply with the protocol for the duration of the study, including hospital visits for treatment and scheduled follow-up visits and examinations.
13. FEV1 ≥ 40% (%Soll)
14. Adequate bone marrow and renal function including the following:

    * Hemoglobin ≥ 9.0 g/dL;
    * Absolute neutrophil count ≥ 1.0 x 10^9/L;
    * Platelets ≥75x 10^9/L;
    * Calculated creatinine clearance ≥30 mL/min as determined by the Cockcroft-Gault equation
15. Adequate hepatic function (with stenting for any obstruction, if required) including the following:

    * Serum bilirubin ≤ 3 x institutional upper limit of normal (ULN);
    * AST (SGOT) / ALT (SGPT) and alkaline phosphatase ≤ 2.5x ULN

    Following exceptions apply:
    * Patients with documented liver metastases: AST and/or ALT ≤ 5x ULN
    * Patients with documented liver or bone metastases: alkaline phosphatase ≤ 5x ULN.
16. Female patients with reproductive potential must have a negative urine or serum pregnancy test within 7 days prior to start of trial.
17. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

    * Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
    * Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).

Exclusion Criteria:

1. Previous treatment with CD137 agonists, immune-checkpoint blockade therapies, anti-PD-1, or anti-PD-L1 therapeutic antibodies (with the exclusion of prior immunotherapy as defined in inclusion criterion 6).
2. Prior therapy for limited-stage SCLC with curative intent.
3. Prior radiotherapy of lung and mediastinal lymph nodes within the past 5 years before the first dose of study drug.
4. Oxygen-dependent medical condition.
5. History or current radiology suggestive of interstitial lung disease (ILD) (including but not limited to idiopathic pulmonary fibrosis (IPF)/usual interstitial pneumonia (UIP)/cryptogenic fibrosing alveolitis (CFA)), non-infectious pneumonitis, drug-induced pneumonitis, idiopathic pneumonitis.
6. Criterion removed.
7. Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study, or during the follow-up period of an interventional study.
8. Participation in another clinical study with an investigational product within 21 days prior to the first dose of the study treatment.
9. Any concurrent chemotherapy, investigational product (IMP), biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer related conditions (e.g., hormone replacement therapy) is acceptable.
10. Major surgery (as defined by the Investigator) within 4 weeks prior to enrollment into the study; patients must have recovered from effects of any major surgery. Note: Local non-major surgery for palliative intent is acceptable.
11. Active or prior documented autoimmune or inflammatory disorders (including but not limited to diverticulitis [with the exception of diverticulosis], celiac disease, systemic lupus erythematosus, Sarcoidosis, or Wegener's syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis). The following are exceptions to this criterion:

    * Patients with vitiligo or alopecia
    * Patients with hypothyroidism (e.g., following Hashimoto's disease) stable on hormone replacement
    * Patients with controlled Type I diabetes mellitus on an insulin regimen
    * Any chronic skin condition that does not require systemic therapy
    * Patients without active disease in the last 5 years may be included but only after consultation with the study physician.
12. Active, uncontrolled inflammatory bowel disease [e.g. ulcerative colitis or Crohn's disease]. Patients in stable remission for more than 1 year may be included.
13. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, uncontrolled cardiac arrhythmia, interstitial lung disease, gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
14. History of another primary malignancy except for:

    * Malignancy treated with curative intent and with no known active disease ≥ 3 years before the first dose of IMP and of low potential risk for recurrence
    * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
    * Adequately treated carcinoma in situ without evidence of disease
15. History of active primary immunodeficiency
16. History of allogenic organ or tissue transplantation.
17. Clinical diagnosis of active tuberculosis.
18. Positive testing for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV RNA) indicating acute or chronic infection. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
19. Positive testing for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
20. Current or prior use of immunosuppressive medication within 14 days before the first dose of atezolizumab. The following are exceptions to this criterion:

    * Intranasal, inhaled, topical steroids, or local steroid injections (e.g. intra articular injection)
    * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
    * Steroids as premedication for hypersensitivity reactions (e.g. CT scan premedication)
21. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 5 months after the last dose of atezolizumab monotherapy.
22. Known allergy or hypersensitivity to the IMP or any of the constituents of the product.
23. Any co-existing medical condition that in the investigator's judgement will substantially increase the risk associated with the patient's participation in the study.
24. Patient who has been incarcerated or involuntarily institutionalized by court order or by the authorities.
25. Patients who are unable to consent because they do not understand the nature, significance and implications of the clinical trial and therefore cannot form a rational intention in the light of the facts.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2024-09-02 (Actual); Study Completion 2024-09-02 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | at 24 month after lat patient randomized
  time from randomization to death

SECONDARY OUTCOMES:
1-year Overall Survival (OS) rate | at 1 year after randomization
  OS rate after 1 year after randomization
2-year Overall Survival (OS) rate | at 2 years after randomization
  OS rate after 2 years after randomization
Progression-free survival (PFS) | at study end (approx. 2 years after last patient randomized)
  PFS is defined as time from randomization to the date of first observed disease progression (investigator assessment according to RECIST 1.1) or death from any cause
objective response rate (ORR) | at study end (approx. 2 years after last patient randomized)
  ORR will be assessed according to RECIST 1.1. The objective response rate will be defined as the proportion of allocated / randomized subjects with best response of complete or partial response.
Intrathoracic tumor control | at study end (approx. 2 years after last patient randomized)
  rate of intrathoracic progression will be determined via assessing the proportion of allocated / randomized subjects with an intrathoracic progression (investigator assessment according to RECIST 1.1).
Incidence, nature, causal relationship and severity of Adverse Events | at study end (approx. 2 years after last patient randomized)
  Incidence, nature, causal relationship and severity of Adverse Events according to CTC v5.0
Frequency of abnormal laboratory parameters | at study end (approx. 2 years after last patient randomized)
  Frequency of abnormal laboratory parameters
frequency of treatment withdrawal | at study end (approx. 2 years after last patient randomized)
  description of relative and absolute frequencies of treatment withdrawal (either due to adverse events or other reasons), which will be compared between treatment groups
completion of radiotherapy | at study end (approx. 2 years after last patient randomized)
  relative and absolute numbers of radiotherapy completers
Cancer related quality of life (Functional Assessment of Cancer Therapy for patients with Lung cancer (FACT-L)) | at study end (approx. 2 years after last patient randomized)
  Cancer-related quality of life measured via the total- and subscores of FACT-L will be compared between the two treatments by analyzing the mean change from baseline. Score scales are ranging from 0 (minimum) to 4 (maximum).

OTHER OUTCOMES:
Collection of biomarker samples for separate biomarker research project | at study end (approx. 2 years after last patient randomized)
  Collection of biomarker samples for separate biomarker research project

CONTACTS AND LOCATIONS:
Overall Officials: Farastuk Bozorgmehr, Dr. med., Principal Investigator — Thoraxklinik at Heidelberg University
Locations (20):
- Austria (2):
  - Klinikum Klagenfurt am Wörthersee, Klagenfurt
  - Kepler Universitätsklinikum, MC III., Pneumologie, Linz
- Germany (18):
  - DRK Kliniken Berlin-Mitte, Berlin
  - Kliniken der Stadt Köln gGmbH Lungenklinik Köln-Merheim, Cologne
  - Universitätsklinikum Carl-Gustav-Carus Dresden, Dresden
  - Universitätsklinikum Essen, Essen
  - Universitätsmedizin Göttingen, Göttingen
  - Medizinische Hochschule Hannover, Hanover
  - Thoraxklinik am Universitätsklinikum Heidelberg, Heidelberg
  - Lungenklinik Hemer, Hemer
  - Klinik Löwenstein gGmbH, Löwenstein
  - Klinikum Ludwigsburg, Ludwigsburg
  - Universitätsmedizin Mainz, Mainz
  - Klinikum der Universität München, München
  - Klinikum Bogenhausen, München
  - Gemeinschaftspraxis für Hämatologie und Onkologie, Münster
  - Sana Klinikum Offenbach GmbH, Offenbach
  - Krankenhaus Barmherzige Brüder, Regensburg
  - Vinzent von Paul Kliniken gGmbH Marienhospital Stuttgart, Stuttgart
  - Universitätsklinikum Ulm, Ulm

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared.

REFERENCES:
- [Derived] Bozorgmehr F, Christopoulos P, Chung I, Cvetkovic J, Feisst M, Krisam J, Schneider MA, Heussel CP, Kreuter M, Muller DW, Thomas M, Rieken S. Protocol of the TREASURE study: Thoracic RadiothErapy with Atezolizumab in Small cell lUng canceR Extensive disease - a randomized, open-label, multicenter phase II trial. BMC Cancer. 2022 Sep 24;22(1):1011. doi: 10.1186/s12885-022-10074-9. PMID 36153496